CLINICAL TRIAL: NCT00911547
Title: A Multicenter, Randomized, Placebo-Controlled, Double-Blind, 2-Period, Parallel-Group Study to Assess the Clinical Effect of MK0476 With Concomitant Administration of and Removal of Inhaled Beclomethasone in Asthmatic Patients
Brief Title: The Clinical Effect of MK0476 With Concomitant Administration of and Removal of Inhaled Beclomethasone in Asthmatic Patients (0476-029)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0476-029; 2009_596
Record Dates: First submitted 2009-05-29; First posted 2009-06-02 (Estimated); Results first posted 2010-06-09 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Asthma
Keywords: chronic asthma
MeSH Terms: conditions — Asthma | interventions — montelukast; Beclomethasone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Experimental): Montelukast + Beclomethasone
  Interventions: Drug: montelukast sodium; Drug: beclomethasone
- 2 (Experimental): Montelukast + Placebo inhaler
  Interventions: Drug: montelukast sodium; Drug: Placebo inhaler
- 3 (Experimental): Placebo tablet + Beclomethasone
  Interventions: Drug: beclomethasone; Drug: placebo tablet
- 4 (Placebo Comparator): Placebo tablet + Placebo inhaler
  Interventions: Drug: Placebo inhaler; Drug: placebo tablet

INTERVENTIONS:
Drug: montelukast sodium — 10 mg tablet taken once daily at bedtime for 16 weeks
  Other Names: MK0476
  Arms: 1; 2
Drug: beclomethasone — 200 ug inhaled, taken twice daily for 16 weeks
  Arms: 1; 3
Drug: Placebo inhaler — placebo inhaler taken twice daily for 16 weeks
  Arms: 2; 4
Drug: placebo tablet — placebo tablet taken once daily at bedtime for 16 weeks
  Arms: 3; 4

SUMMARY:
This study will investigate the additive effect of montelukast (MK0476) taken along with inhaled beclomethasone versus inhaled beclomethasone alone.

ELIGIBILITY:
Inclusion Criteria:

* Female patients tested negative for pregnancy and agreed to use appropriate contraceptives through out the study
* Patient was a nonsmoker
* Patient was in good general health (except for asthma)

Exclusion Criteria:

* Patient was hospitalized
* Patient was female who was less than 8 weeks postpartum or breast feeding
* Patient planned to move or vacation away during the study
* Patient had major surgery within 4 weeks the past 4 weeks
* Patient has donated blood or participated in a clinical trial within the past 4 weeks
* Patient was a regular user or recent abuser of alcohol or illicit drugs
* Patient was 40% over or under normal weight for height

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 642 (Actual)
Dates: Start 1995-03; Primary Completion 1996-04 (Actual); Study Completion 1996-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Laviolette M, Malmstrom K, Lu S, Chervinsky P, Pujet JC, Peszek I, Zhang J, Reiss TF. Montelukast added to inhaled beclomethasone in treatment of asthma. Montelukast/Beclomethasone Additivity Group. Am J Respir Crit Care Med. 1999 Dec;160(6):1862-8. doi: 10.1164/ajrccm.160.6.9803042. PMID 10588598

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at 22 sites in the United States (US) and 48 sites in 16 other countries in North America, Europe, Africa, Australia, and Southeast Asia.
  Publication incorrectly listed 18 participating countries. Results posting is correct with 17 countries.
  Prime therapy period: March 1995 to April 1996.
Pre-assignment Details: Patients received inhaled beclomethasone (200 μg twice daily) starting at the Prestudy Visit and continuing through the single-blind run-in period. Patients who experienced worsening asthma requiring more than albuterol therapy (inhaled or nebulized) did not qualify for randomization.
Groups:
- Placebo: Montelukast (MK) placebo tablet orally once daily at bedtime. Beclomethasone (beclo) inhaler was removed in a blinded, two-step procedure over 4 weeks (wks): beclomethasone inhaler 4 puffs (50 μg/puff) upon arising (Weeks 1 to 2)) and 4 puffs (50 μg/puff) at bedtime (Weeks 1 to 4); beclomethasone placebo inhaler 4 puffs upon arising (Weeks 3 to 16) and 4 puffs at bedtime (Weeks 5 to 16). Albuterol inhaler as needed.
- Montelukast: MK 10 mg tablet orally once daily at bedtime. Beclomethasone was removed in a blinded, two-step procedure over 4 weeks: beclomethasone inhaler 4 puffs (50 μg/puff) upon arising (Weeks 1 to 2) and 4 puffs (50 μg/puff) at bedtime (Weeks 1 to 4); beclomethasone placebo inhaler 4 puffs upon arising (Weeks 3 to 16) and 4 puffs at bedtime (Weeks 5 to 16). Albuterol inhaler as needed.
- Beclomethasone: MK placebo tablet orally once daily at bedtime and beclomethasone inhaler 4 puffs (50 μg/puff) upon arising and 4 puffs (50 μg/puff) at bedtime for 16 Weeks. Albuterol inhaler as needed.
- Montelukast+ Beclomethasone: MK 10 mg tablet orally once daily at bedtime and beclomethasone inhaler 4 puffs (50 μg/puff) upon arising and 4 puffs (50 μg/puff) at bedtime for 16 Weeks. Albuterol inhaler as needed.
Period: Overall Study
Arm/Group | Placebo | Montelukast | Beclomethasone | Montelukast+ Beclomethasone
Started | 48 (Efficacy in last 10 wks to minimize confounding effect of beclo in 1st 4 wks & allow beclo washout.) | 201 (Efficacy in last 10 wks to minimize confounding effect of beclo in 1st 4 wks & allow beclo washout.) | 200 (Efficacy analyses were over the 16 weeks of treatment.) | 193 (Efficacy analyses were over the 16 weeks of treatment.)
Completed | 37 | 159 | 178 | 177
Not Completed | 11 | 42 | 22 | 16
Not completed — Adverse Event | 8 | 27 | 11 | 6
Not completed — Lost to Follow-up | 0 | 0 | 2 | 1
Not completed — Protocol Violation | 0 | 5 | 5 | 1
Not completed — Withdrawal by Subject | 3 | 10 | 4 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Montelukast | Beclomethasone | Montelukast+ Beclomethasone | Total
Number analyzed (Participants) | 48 | 201 | 200 | 193 | 642
Age, Continuous [Mean (Full Range); unit: years] | 40.50 [15 to 75] | 38.00 [15 to 75] | 39.00 [15 to 78] | 40.00 [15 to 76] | 39.00 [15 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 102 | 96 | 85 | 312
  Male | 19 | 99 | 104 | 108 | 330
Race/Ethnicity [Number; unit: participants]
  Caucasian | 40 | 189 | 184 | 177 | 590
  Black | 4 | 3 | 4 | 5 | 16
  Hispanic | 2 | 5 | 1 | 6 | 14
  Other | 2 | 4 | 11 | 5 | 22
Daytime symptom score [Mean (Standard Deviation); unit: Units on a Scale] — Daytime symptom score: The patient scored his/her symptoms [from 0
  (best) to 6 (worst)] on a daily basis.
  Units on a Scale | 2.36 (0.68) | 2.14 (0.83) | 2.17 (0.82) | 2.17 (0.84) | 2.18 (0.82)
Forced expiratory volume in 1 second (FEV1) [Mean (Standard Deviation); unit: Liters] | 2.45 (0.69) | 2.61 (0.74) | 2.53 (0.68) | 2.61 (0.68) | 2.57 (0.70)
Morning peak flow rate (PEFR) [Mean (Standard Deviation); unit: Liters/minute] | 406.80 (73.47) | 419.94 (92.47) | 402.91 (86.19) | 412.46 (91.15) | 411.42 (88.92)
Nocturnal asthma score [Mean (Standard Deviation); unit: Units on a Scale] — Nocturnal asthma score: The patient scored his/her symptoms [from 0 (best)
  to 3 (worst)] on a daily basis.
  Units on a Scale | 0.57 (0.46) | 0.41 (0.45) | 0.35 (0.44) | 0.43 (0.47) | 0.41 (0.46)
Total daily Beta-agonist use [Mean (Standard Deviation); unit: Puffs] — Number of inhalations (Puffs) of beta-agonist medication
  Puffs | 4.16 (3.02) | 3.52 (2.34) | 3.51 (2.47) | 3.41 (2.17) | 3.53 (2.39)

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) in Patients With Chronic Asthma
Description: Mean percent change from baseline in FEV1 in patients with chronic asthma averaged over 16 weeks for the Beclo and MK+ Beclo groups and averaged over last 10 weeks for the Placebo and MK groups
Time Frame: Baseline & over 16 weeks for the Beclomethasone (Beclo) and Montelukast (MK) + Beclo groups and over last 10 weeks for the Placebo and MK groups
Population: Primary efficacy analyses were based on the intention-to-treat principle, i.e., inclusion of all patients with a baseline and at least one postbaseline measurement. No missing values were imputed. Data collected during discontinuation and unscheduled visits were included the analysis. Differences between treatments are evaluated based on LS means
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of Change
Arm/Group | Placebo | Montelukast | Beclomethasone | Montelukast+ Beclomethasone
Number analyzed (Participants) | 44 | 183 | 198 | 191
Percentage of Change | -11.96 [-16.28 to -7.64] | -5.31 [-7.32 to -3.30] | 0.72 [-0.89 to 2.33] | 5.08 [3.43 to 6.74]

2. Primary Outcome: Mean Change From Baseline in Daytime Symptom Score on the Daytime Asthma Symptoms Diary in Patients With Chronic Asthma
Description: The daily daytime symptom score was determined by averaging the daily scores (the patient scored his/her symptoms [from 0 (best) to 6 (worst)] on a daily basis.) for the four questions on the Daytime Asthma Symptoms Diary.
  The average daytime symptom score for the visit was determined by averaging the daily symptom scores over all days between two consecutive visits.
Time Frame: Baseline & over 16 weeks for the Beclo and MK + Beclo groups and over last 10 weeks for the Placebo and MK groups
Population: Primary efficacy analyses were based on the intention-to-treat principle, i.e., inclusion of all patients with a baseline and at least one postbaseline measurement. No missing values for this analysis were imputed. Data collected during discontinuation visits and unscheduled visits were included in this analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Montelukast | Beclomethasone | Montelukast+ Beclomethasone
Number analyzed (Participants) | 44 | 183 | 198 | 191
Units on a Scale | 0.31 [0.08 to 0.54] | 0.27 [0.17 to 0.38] | -0.02 [-0.10 to 0.06] | -0.13 [-0.22 to -0.05]

3. Secondary Outcome: Mean Percent Change From Baseline in Total Daily Beta-agonist Medication Use
Description: Beta-agonist medication use from the daytime and overnight asthma symptoms diaries for each 24-hour period was added to determine the daily total number of puffs used. The average daily number of puffs for the visit was determined as the average daily number of puffs over all days between consecutive visits.
Time Frame: Baseline & over 16 weeks for the Beclo and MK + Beclo groups and over last 10 weeks for the Placebo and MK groups
Population: Efficacy analyses were based on the intention-to-treat principle, i.e., inclusion of all patients with a baseline and at least one postbaseline measurement. No missing values for this analysis were imputed. Data collected during discontinuation visits and unscheduled visits were included in this analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Montelukast | Beclomethasone | Montelukast+ Beclomethasone
Number analyzed (Participants) | 44 | 180 | 194 | 189
Percent Change | 59.20 [25.77 to 92.63] | 44.48 [28.82 to 60.14] | 6.04 [-3.78 to 15.86] | -5.51 [-15.54 to 4.52]

4. Secondary Outcome: Mean Change From Baseline in Morning Peak Flow Rate (PEFR) in Patients With Chronic Asthma
Description: Morning PEFR was measured in triplicate immediately upon arising before taking any medication and the best value recorded on the overnight asthma symptoms diary. The mean morning PEFR for the visit was determined by averaging all valid PEFR measurements for the days between consecutive visits.
Time Frame: Baseline & over 16 weeks for the Beclo and MK + Beclo groups and over last 10 weeks for the Placebo and MK groups
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters/minute
Arm/Group | Placebo | Montelukast | Beclomethasone | Montelukast+ Beclomethasone
Number analyzed (Participants) | 44 | 184 | 197 | 191
Liters/minute | -27.10 [-38.96 to -15.25] | -15.37 [-20.87 to -9.87] | 2.65 [-1.31 to 6.60] | 10.41 [6.36 to 14.47]

5. Secondary Outcome: Mean Change From Baseline in Nocturnal Asthma Score on the Overnight Asthma Symptoms Diary in Nocturnal Asthmatic Patients Only
Description: Mean change from baseline in Nocturnal asthma score; the patient scored his/her symptoms [from 0 (best) to 3 (worst)] on a daily basis. Responses to the question, "Did you wake up with asthma symptoms?" (no, once, more than once, awake "all night"), were assigned numerical values (0, 1, 2, 3, respectively).
  The average score for the visit was determined by averaging the daily scores over all days between consecutive visits.
Time Frame: Baseline & over 16 weeks for the Beclo and MK + Beclo groups and over last 10 weeks for the Placebo and MK groups
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Montelukast | Beclomethasone | Montelukast+ Beclomethasone
Number analyzed (Participants) | 27 | 84 | 74 | 85
Units on a Scale | 0.17 [-0.01 to 0.35] | 0.18 [0.09 to 0.28] | -0.06 [-0.14 to 0.02] | -0.20 [-0.28 to -0.12]

ADVERSE EVENTS:
Time Frame: Over 16 weeks of treatment and for 14 days post-treatment
Arm/Group | Placebo | Montelukast | Beclomethasone | Montelukast+ Beclomethasone
Serious Adverse Events (participants affected / at risk) | 1/48 | 4/201 | 6/200 | 1/193
Other Adverse Events (participants affected / at risk) | 36/48 | 150/201 | 139/200 | 123/193
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=48) | Montelukast (N=201) | Beclomethasone (N=200) | Montelukast+ Beclomethasone (N=193)
Fracture, Ankle (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Pain, Back (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Neurological Disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 2 | 0
Surgery, Nasopharyngeal (Surgical and medical procedures) | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=48) | Montelukast (N=201) | Beclomethasone (N=200) | Montelukast+ Beclomethasone (N=193)
Asthenia/Fatigue (General disorders) | 3 | 2 | 1 | 3
Pain, Abdominal (General disorders) | 0 | 4 | 7 | 10
Nausea (Gastrointestinal disorders) | 0 | 12 | 11 | 5
Pain, Back (Musculoskeletal and connective tissue disorders) | 2 | 9 | 6 | 10
Headache (Nervous system disorders) | 6 | 52 | 42 | 50
Asthma (Respiratory, thoracic and mediastinal disorders) | 20 | 75 | 40 | 23
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 4 | 7 | 4 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 11 | 5 | 8
Infection, Respiratory, Upper (Infections and infestations) | 19 | 72 | 79 | 70
Influenza (Infections and infestations) | 3 | 15 | 11 | 11
Pharyngitis (Infections and infestations) | 2 | 12 | 16 | 10
Sinusitis (Infections and infestations) | 2 | 12 | 9 | 8
Rash (Skin and subcutaneous tissue disorders) | 3 | 7 | 3 | 1

LIMITATIONS AND CAVEATS:
Efficacy over 16 weeks of treatment for Beclo and MK+Beclo groups, and last 10 weeks for Placebo and MK groups to minimize confounding effect of beclo in 1st 4 weeks of treatment and to allow beclo washout.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.